CLINICAL TRIAL: NCT04898569
Title: Effect of Intravenous Ferric Carboxymaltose on Hemoglobin Response and Transfusion in Patients With Iron Deficiency Anemia After Off-Pump Coronary Artery Bypass Grafting
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2018-0371
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Coronary Artery Disease
Keywords: Bleeding; Blood transfusion; Coronary artery bypass surgery; Hemostasis; Iron therapy
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: In cardiac surgery, patients were randomized to receive Ferinject or placebo (n=50), respectively. The selected agent was intravenous infusion in general ward, preoperatively.
Who Masked: Participant
Masking Description: Patients were offered the allocated treatment for ferric carboxymaltose or not, using the block randomization system. The selected agent was infused to patients after randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferinject® (Experimental)
  Interventions: Drug: Ferinject
- Normal saline (Placebo Comparator)
  Interventions: Drug: Normal Saline Flush

INTERVENTIONS:
Drug: Ferinject — Ferric carboxymaltose injection
  Other Names: Colloidal solution of the iron complex ferric carboxymaltose
  Arms: Ferinject®
Drug: Normal Saline Flush — placebo
  Other Names: placebo comparator
  Arms: Normal saline

SUMMARY:
In this prospective open-label randomized tral, 100 patients with elective off-pump coronary artery bypass (OPCAB) or minimal invasive direct coronary bypass (MIDCAB) surgery were enrolled. Before surgery, if a patient had iron deficiency anemia, the patient was randomized to receive Ferinject®(Ferric carboxymaltose, n=50) or placebo (normal saline, n=50), respectively. A single dose should not exceed 1000mg of iron per day or 20mg per kg body weight. In addition, the administration of 1000mg of iron should not exceed once a week. Administration to patients with hemodialysis-dependent chronic kidney disease is once daily, and the maximum dose should not exceed 200 mg (4 ml) of iron. Patients weighing less than 35 kg should not exceed 500 mg total iron dose. It uses intravenous infusion and can be administered up to 1,000mg (20ml) as the maximum iron once. For intravenous infusion, this drug is diluted with 0.9% sterile physiological saline solution.

DETAILED DESCRIPTION:
* Perioperative blood loss and iatrogenic hemodilution lead to postoperative anemia which correlates with infections, and poor physical function, mobility and recovery with subsequent increases in the length of hospital stay and mortality. Preoperative anemia management reduce intraoperative blood loss such as normothermia, antifibrinolytics and cell salvage are key strategies to ameliorate postoperative anemia.
* Patient screening method Off-pump coronary artery bypass (OPCAB) under median-sternotomy, or minimal invasive direct coronary bypass (MIDCAB) undertaken under median-sternotomy Among them, the selection/exclusion criteria are checked and the subjects of the study are screened. * Inclusion/ exclusion criteria **Inclusion:

  * Patients with Preoperative iron deficiency anemia Among Patients scheduled for cardiopulmonary coronary artery bypass graft under median sternotomy in cardiovascular surgery **Exclusion: - a) Patients who underwent iron correction treatment (oral, injection, blood transfusion) within 2 months prior to surgery b) Patients taking anticoagulants before surgery c) Patients taking and administering drugs that can cause bone marrow suppression, such as anticancer drugs, before surgery d) Patients with chronic liver disease and chronic kidney disease undergoing dialysis e) Patients scheduled for coronary artery bypass graft for emergency surgery f) Patients with a history of hypersensitivity reactions and side effects to iron drugs g) Minor (under 20 years old) 3) Definition of iron deficiency anemia (if all criteria a to c in the following items are satisfied)

    1. Ferritin<300mcg/L
    2. Transferrin saturation<25%
    3. Hb<12.0g/dL for women or Hb<13.0g/dL for men * The primary goal of this study was the effect of intravenous administration of ferric carboxymaltose on postoperative hemoglobin levels in patients with preoperative iron deficiency anemia among patients requiring cardiopulmonary coronary artery bypass grafting due to coronary artery disease. It is to analyze the effect compared to the control.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 19 years or older
2. undergoing elective OPCAB or MIDCAB surgery with multi-vessel coronary artery disease.

Exclusion Criteria:

1. Patients who underwent iron correction treatment (oral, injection, blood transfusion) within 2 months prior to surgery
2. Patients taking anticoagulants before surgery
3. Patients taking and administering drugs that can cause bone marrow suppression, such as anticancer drugs, before surgery
4. Patients with chronic liver disease and chronic kidney disease undergoing dialysis
5. Patients scheduled for coronary artery bypass graft for emergency surgery
6. Patients with a history of hypersensitivity reactions and side effects to iron drugs
7. Minor (under 20 years old)
8. Definition of iron deficiency anemia (if all criteria a to c in the following items are satisfied)

   1. Ferritin<300mcg/L
   2. Transferrin saturation<25%
   3. Hb<12.0g/dL for women or Hb<13.0g/dL for men

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Total mediastinal blood loss and transfusion counts | At admission periods for Off-Pump Coronary Artery Bypass or Minimally Invasive Direct Coronary Artery Bypass surgery (Mean 8~9 days)
  For cost-effectiveness analysis of ferric carboxymaltose in preoperative iron treatment

SECONDARY OUTCOMES:
blood loss in the operative day | 24 hours later after surgery
amount of blood products transfused both intraoperatively and postoperatively | 24 hours later after surgery
rate of surgical revision for bleeding | intraoperative
total length of intensive care unit (ICU) stay | mean 3-4 days
rate of postoperative morbidity | Participants will be followed during 1 years from operation
rate of postoperative mortality | Participants will be followed during 1 years from operation

CONTACTS AND LOCATIONS:
Overall Officials: Young-Nam Youn, Principal Investigator — Division of Cardiovascular Surgery, Severance Cardiovascular Hospital, Yonsei University College of Medicine
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banerjee S, McCormack S. Intravenous Iron Preparations for Patients Undergoing Elective Surgery: A Review of Clinical Effectiveness, Cost-Effectiveness, and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2019 Mar 27. Available from http://www.ncbi.nlm.nih.gov/books/NBK545893/ PMID 31487129